CLINICAL TRIAL: NCT06898970
Title: An Open-Label, Multicenter, Phase 2 Study With Safety Lead-In of Intratumoral Vusolimogene Oderparepvec (VO) in Combination With Pembrolizumab in Patients With Angiosarcoma
Brief Title: Intratumoral Vusolimogene Oderparepvec (VO) in Combination With Pembrolizumab for Angiosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Varun Monga, MBBS (Other)
Collaborators: Replimune Inc. (Industry)
Responsible Party: Sponsor-Investigator, Varun Monga, MBBS, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25871; NCI-2025-02056 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Angiosarcoma; Angiosarcoma, Adult
Keywords: Immunotherapy
MeSH Terms: conditions — Hemangiosarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Vusolimogene Oderparepvec (VO), Pembrolizumab) (Experimental): All participants receive a single dose of VO on Day -14. On Cycle 1 Day 1 (C1D1), participants receive second dose of VO, and subsequent doses occur every 3 weeks for 7 cycles in combination with 200 mg pembrolizumab every 3 weeks for 8 cycles starting C1D1. After 8 cycles of pembrolizumab, participants may have the pembrolizumab dose schedule altered to a single 400 mg dose every 6 weeks, and treatment with pembrolizumab may continue for up to 2 years after starting first dose on C1D1. Participants may receive up to eight additional doses of VO after progression for a total of 16 dosing days. Safety follow up visits occur 30 and 90 days after last dose of either treatment (whichever drug was taken last) or after the participant has taken 2 years of pembrolizumab as a part of this study.
  Interventions: Biological: Vusolimogene Oderparepvec (VO); Drug: Pembrolizumab

INTERVENTIONS:
Biological: Vusolimogene Oderparepvec (VO) — Given intratumorally
  Other Names: RP1
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda

SUMMARY:
This is a multicenter, open-label study of Intratumoral Vusolimogene Oderparepvec (VO) to investigate safety and estimate when used in combination with pembrolizumab for treating participants with angiosarcoma. This is the first study evaluating this novel combination in participants with advanced angiosarcoma who have progressed after prior immunotherapy.

DETAILED DESCRIPTION:
Primary Objectives:

Safety Lead-in:

I. To assess the safety and tolerability of VO in combination with pembrolizumab.

Phase 2:

1. To assess the efficacy of VO in combination with pembrolizumab as determined by objective response rate (ORR).
2. To assess the safety and tolerability of VO in combination with pembrolizumab.

Secondary Objectives:

1. To assess the duration of response (DOR).
2. To assess the complete response rate (CRR), clinical benefit rate (CBR), progression free survival, and 1-year and 2-year overall survival (OS).
3. To further assess the efficacy of VO in combination with pembrolizumab as determined by objective response rate (ORR) per modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

OUTLINE:

Participants may continue study treatment for up to 2 years with pembrolizumab and 24 weeks with VO. Some participants may be eligible to receive treatment after progression. For participants who discontinued for reasons other than confirmed progressive disease (PD) or completed treatment, tumor response assessments will continue approximately every 12 weeks from the last tumor assessment for up to two years or until the start of subsequent anticancer treatment, confirmed disease progression, withdrawal of consent, loss to follow-up, death, whichever occurs first. Participants will also be followed-up every 6 months to assess for survival/disease/anti-cancer therapy status for up to 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Participants with biopsy proven cutaneous angiosarcoma that is locally advanced and unresectable or metastatic and has received and progressed on at least one prior immunotherapy based regimen within 6 months prior to screening.
2. At least one measurable tumor of ≥ 1 cm in longest diameter or ≥ 1.5 cm in shortest diameter (for lymph nodes) and injectable lesions which in aggregate comprise >= 1 cm in longest diameter.
3. Participants must have received and progressed following first-line standard of care, including a taxane or anthracycline based chemotherapy regimen.
4. Measurable disease based upon Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Life expectancy of at least 3 months, in the opinion of the treating investigator.
6. Females of childbearing potential must have a negative beta-human chorionic gonadotropin (beta-hCG) test at screening within 7 days of Cycle 1 Day 1.
7. Female participants of reproductive potential must agree to avoid becoming pregnant and adhere to a highly effective contraception method until 90 days after last dose of VO alone or 120 days after last dose of VO and pembrolizumab.
8. Male participants of reproductive potential must agree to avoid impregnating a partner and adhere to a highly effective contraception method until 90 days after last dose of VO study agent and refrain from donating sperm during this period.
9. Age <=18 years on the day of signed informed consent.
10. Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky ≥ 70%)
11. Adequate hematologic function including:

    1. White blood cell count (WBC) >= 2.0 × 109/L
    2. Absolute neutrophil count (ANC) >= 1.5 × 109/L
    3. Platelet count >=100 × 109/L
    4. Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within 2 weeks of dosing)
12. Adequate hepatic function including:

    1. Adequate renal function: Total bilirubin <= 1.5 × upper limit of normal (ULN) (except participants with Gilbert Syndrome who must have a total bilirubin of < 3.0 × ULN) or direct bilirubin <=ULN for a participant with total bilirubin level > 1.5 × ULN. If total bilirubin is > 1.5 × ULN but <= 3 × ULN, both aminotransferase (AST and ALT) levels must be <= 3 × ULN.
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3.0 × ULN (or <= 5.0 × ULN, if liver metastases) Note: If aminotransferase levels (AST and/or ALT) are > 3 × ULN but <= 5 × ULN, total bilirubin must be <= 1.5 × ULN.
    3. Alkaline phosphatase (ALP) <= 2.5 × ULN (or <= 5.0 × ULN, if liver or bone metastases)
13. Blood creatinine <= 1.5 × ULN or measured or calculated (using Cockcroft) creatinine clearance >= 30 mL/minute for participants with creatinine levels > 1.5 × institutional ULN.
14. Adequate coagulation: Prothrombin time (PT) or international normalization ratio (INR) <=1.5 × ULN, and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) <= 1.5 × ULN. Note: For participants who are on chronic anticoagulant therapy these participants may be enrolled if the pretreatment INR < 2.5.
15. Adequate oxygen saturation: >=92% on room air.
16. Ability to understand and the willingness to sign a written informed consent document.
17. Participants with a history of treated brain metastasis and, at the time of screening, asymptomatic CNS metastases are eligible, provided they meet all the following:

    1. Brain imaging at screening shows no evidence of interim progression for at least 4 weeks by repeat imaging, and clinically stable for at least 2 weeks
    2. Have measurable disease outside the central nervous system (CNS)
    3. Only supratentorial metastases allowed
    4. No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
    5. No stereotactic or whole brain radiation within 14 days prior to C1D1.
18. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

1. Prior treatment with an oncolytic therapy.
2. Currently receiving antiviral drug therapy (e.g. valacyclovir or acyclovir).
3. Has acute or chronic active hepatitis B and C virus infection or known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV RNA [qualitative]) or HIV infection.Note: No testing for Hepatitis B, Hepatitis C, or HIV is required unless mandated by local health authority or if clinically indicated.
4. Had systemic infection requiring IV antibiotics or other serious infection within 14 days prior to dosing.
5. Has active significant herpetic infections or prior complications of herpes simplex 1 (HSV-1) infection (e.g., herpetic keratitis or encephalitis).
6. Systemic anticancer therapy within 4 weeks prior to enrollment or five half-lives, whichever is shorter, before the first administration of VO. Note: programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PD-L1) directed therapy is allowed.
7. Has not recovered from adverse events due to prior anti-cancer therapy to <= grade 1 or baseline. Note: participants with toxicities after prior anticancer therapies that are not considered a likely safety risk such as Grade ≤ 2 neuropathy or alopecia, or immune mediated AEs that are unlikely to recur with standard countermeasures (e.g., hormone replacement after adrenal crisis, stable endocrine insufficiencies such as thyroid and adrenal insufficiency), are an exception to this criterion and may qualify for the study in discussion with the Principal Investigator.
8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within four weeks prior to the first dose of study treatment. Note: participants who have entered the follow-up phase of an investigational study may participate as long as it has been four weeks since the last dose of the previous investigational agent.
9. Has received prior radiotherapy within two weeks of start of study treatment. Note: participants who are eligible must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (<=2 weeks of radiotherapy) to non-CNS disease.
10. History of interstitial lung disease.
11. History of documented allergic reactions or acute hypersensitivity attributed to VO and pembrolizumab or any of its excipients.
12. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guérin (BCG), and typhoid vaccine. Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed, however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Available Coronavirus disease of 2019 (COVID-19) vaccines do not contain live virus and are allowed.
13. Conditions requiring treatment with immunosuppressive doses (> 10 mg daily prednisone or equivalent) of systemic corticosteroids other than for corticosteroid replacement therapy within 14 days after enrollment. For the definition of replacement therapy.
14. Undergo major surgery ≤ 2 weeks prior to starting VO. Note: participants who undergo major surgery requiring general anesthesia such as exploratory laparotomy or thoracotomy and are eligible for the study must adequately recover prior to starting study treatment. Procedures such as central line placement, endoscopies and tooth extractions under local anesthesia do not meet criteria for major surgery.
15. Has a history of (non-infectious) pneumonitis that required corticosteroids or has current pneumonitis.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs, or interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
17. Has known psychiatric, alcohol abuse, or substance abuse disorders that would interfere with cooperating with the requirements of the study.
18. Has serious uncontrolled medical disorders such as uncontrolled hypertension, bleeding diatheses, uncontrolled diabetes.
19. Has clinically significant cardiovascular disease within 12 months from first dose of study drug, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, history of myocarditis, or cardiac arrhythmia associated with hemodynamic instability.
20. Is a person deprived of their liberty by a judicial or administrative decision, or an adult person subject to a legal protection measure.
21. Has been treated with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to first dose and throughout the study.
22. Has an active, known, or suspected autoimmune disease. Note: participants with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
23. Has a history of life-threatening toxicity related to prior immune therapy. Note: Toxicities that are unlikely to recur with standard countermeasures (e.g., hormone replacement after adrenal crisis) are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with reported treatment-emergent adverse events (Safety Lead-In) | Up to 1 year
  Safety and tolerability will be reported as the percentage of the first 6 participants (the safety-lead in participants) who received at least one dose of study treatment with any reported treatment-emergent adverse events (TEAEs), >= Grade 3 TEAEs, serious adverse events (SAEs), and TEAEs requiring discontinuation of VO. Adverse events will be classified using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Proportion of participants who experience an objective response (Phase 2 participants) | Up to 1 year
  Objective response will be measured per RECIST v. 1.1 and is defined as complete response (CR) or partial response (PR) and confirmed by repeat imaging >=4 weeks after assessment for participants who completed at least 4 of the planned 8 intratumoral injections.
Percentage of participants with reported treatment-emergent adverse events | Up to 1 year
  The percentage of all participants who received at least one dose of study treatment with any treatment-emergent adverse events (TEAEs), ≥ Grade 3 TEAEs, serious adverse events (SAEs), and TEAEs requiring discontinuation of VO. Adverse events will be classified using NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0.

SECONDARY OUTCOMES:
Median Duration of Response (DOR) | Up to 1 year
  The DOR is the time from the first day of documented response until disease progression. Objective response will be measured per RECIST v. 1.1 and is defined as complete response (CR), partial response (PR), or stable disease (SD) and confirmed by repeat imaging >=4 weeks after assessment for participants who completed at least 4 of the planned 8 intratumoral injections. The median time in months will be reported along with 25% confidence intervals.
Percentage of participants with documented Complete Response (CRR) | Up to 1 year
  The CRR is the percentage of participants with a demonstrated complete response as measured per RECIST v. 1.1 and confirmed by repeat imaging >=4 weeks after assessment for participants who completed at least 4 of the planned 8 intratumoral injections will be reported
Percentage of participants with documented Clinical Benefit (CBR) | Up to 1 year
  The percentage of participants with demonstrated Clinical Benefit as measured per modified RECIST v. 1.1 criteria and is defined as having a complete response (CR), partial response (PR), or stable disease (SD) and confirmed by repeat imaging >=4 weeks after assessment for participants who completed at least 4 of the planned 8 intratumoral injections for greater than 3 months (>=4 months)
Median Progression-Free Survival (PFS) | Up to 2 years
  The time that elapses between Day -14 and the earlier of the day of first documented disease progression or death from any cause for all evaluable patients. Disease progression is defined as progressive disease (PD) per modified RECIST 1.1,1 other documented clinical or radiographical progression per physician judgement, or death due to disease.
Median Overall Survival | Up to 2 years
  The OS is defined as the time that elapses in months between Day -14 and the date of death from any cause for all participants.
Percentage of participants who experience an objective response | Up to 1 year
  Objective response will be measured per RECIST v. 1.1 and is defined as complete response (CR) or partial response (PR) and confirmed by repeat imaging >=4 weeks after assessment for participants who completed at least 4 of the planned 8 intratumoral injections and will be collected up to 30 days after the last dose of either study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Varun Monga, MBBS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets may be shared with study collaborators during the course of the study through study closure.
Supporting Information: Study Protocol, SAP, ICF